CLINICAL TRIAL: NCT03543228
Title: Prefect Study of MyoStrain CMR for the Detection of Cardiotoxicity
Brief Title: MyoStrain CMR for the Detection of Cardiotoxicity
Acronym: Prefect
Status: Completed | Type: Observational
Sponsor: Myocardial Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: VAL-1005P(A)
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cardiotoxicity; Heart Failure; Chemotherapeutic Toxicity
Keywords: Strain
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- MyoStrain: During standard chemotherapy and/or targeted treatment for breast cancer or lymphoma, MyoStrain will be used during standard cardiac magnetic resonance imaging to evaluate the change in myocardial contraction regionally and globally to detect cardiotoxicity and management of myocardial dysfunction.
  Interventions: Diagnostic Test: MyoStrain

INTERVENTIONS:
Diagnostic Test: MyoStrain — MyoStrain quantifies myocardial contraction to detect changes in heart function during chemotherapy.

SUMMARY:
The Prefect Pilot Study evaluates the use of the EC approved MyoStrain SENC CMR Imaging System to detect cardiotoxicity from drugs used to treat cancer (e.g. Breast Cancer and Lymphomas).

DETAILED DESCRIPTION:
The study is a prospective, observational, single center, observational clinical study that will enroll up to 50 patients undergoing chemotherapy and/or targeted therapy with or without concomitant radiotherapy for the treatment of breast cancer or lymphoma. Enrolled subjects will be evaluated with the MyoStrain SENC CMR Imaging System that measures myocardial strain during standard Cardiac Magnetic Resonance imaging at baseline through 6 month follow-up.

The MyoStrain SENC CMR Imaging System has been approved with an EC Certificate according to Directive 93/42/EEC on Medical Devices, Annex II excluding Section 4 (CE 657862) in respect of: Design, development and manufacture of software for the quantification of cardiac MRI images. MyoStrain measures the contraction of heart muscle in one heartbeat per image plane. With 6 image planes (3 short axis & 3 long axis), a complete measure of the health of the myocardium, both regionally and globally, can be obtained within a minute without requiring contrast injection or a breath-hold.

Heart health will be monitored throughout cancer therapy to quantify the toxic effects of chemotherapy with or without a reduction in traditional measures such as ejection fraction, and the ability to reverse observed cardiotoxicity with standard heart failure therapy.

The goal of the study is to determine the ability to detect subclinical cardiotoxicity before extensive damage causes the reduction in traditional measures, which are currently used to categorize heart failure and serve as the basis of treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Chemotherapy for Cancer Treatment
* Provided Written Informed Consent

Exclusion Criteria:

* Contraindication to Magnetic Resonance Imaging
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be carefully selected from the pool of patients currently undergoing or scheduled to undergo chemotherapy for cancer treatment including breast cancer and lymphoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of MyoStrain to Detect Cardiotoxicity | 6 months
  Sensitivity of MyoStrain CMR Software to quantify myocardial dysfunction before changes in traditional measures including ejection fraction as ascertained by Biomarkers including BNP, Troponin, and SF-36 Quality of Life. Sensitivity will be calculated by looking at paired t-test evaluations comparing follow-up time points to baseline as to whether changes associated with administration of chemotherapy agents and/or heart failure therapy are detected.

SECONDARY OUTCOMES:
Cardiotoxicity Incidence of Chemotherapy Drugs | 6 months
  Incidence of subclinical dysfunction during chemotherapy as determined by CMR detection of the amount and locations of declining segmental myocardial contraction with MyoStrain software that measured the ability of the myocardium to contract in 37 segments of the heart (16 longitudinal strain measurements from 3 short axis planes & 21 circumferential strain segments from 3 long-axis planes).
Efficacy of Heart Failure Therapy to Treat Cardiotoxicity | 6 months
  Impact of heart failure medications to improve subclinical dysfunction, calculated by improvement in previously worsened segmental myocardial contraction with MyoStrain software that measured the ability of the myocardium to contract in 37 segments of the heart (16 longitudinal strain measurements from 3 short axis planes & 21 circumferential strain segments from 3 long-axis planes).
Cardiotoxicity Risk Stratification | 6 months
  Ability to detect risk of developing cardiotoxicity by quantifying subclinical myocardial dysfunction in patients with segmental strain at baseline exceeding predefined thresholds. Higher risk patients will be defined as 2 or more segments > -10% with MyoStrain measurements OR 9 or more segments > -17%; Lower risk patients will be the remaining patients. The changes in strain for each patient category will be evaluated by changes in segmental strain during oncology therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Steen, MD, Principal Investigator — Marien Krankenhaus
Locations (1):
- Marien Krankenhaus GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Giusca S, Korosoglou G, Montenbruck M, Gersak B, Schwarz AK, Esch S, Kelle S, Wulfing P, Dent S, Lenihan D, Steen H. Multiparametric Early Detection and Prediction of Cardiotoxicity Using Myocardial Strain, T1 and T2 Mapping, and Biochemical Markers: A Longitudinal Cardiac Resonance Imaging Study During 2 Years of Follow-Up. Circ Cardiovasc Imaging. 2021 Jun;14(6):e012459. doi: 10.1161/CIRCIMAGING.121.012459. Epub 2021 Jun 15. PMID 34126756